CLINICAL TRIAL: NCT02646696
Title: Reliability of Electrodermal Activity: Quantifying Sensory Processing in Children With Autism Spectrum Disorder
Brief Title: Reliability Study Using Electrodermal Activity to Measure Sensory Processing in Children With and Without Autism Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: Barpak Geriatric Health Services, Inc. d/b/a Barpak Occupational Therapy (Other)
Responsible Party: Sponsor
Other Study IDs: Barpak-01-EDA
Record Dates: First submitted 2016-01-04; First posted 2016-01-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children with Autism Spectrum Disorder: Boys between the age of 4 to 11 years old with Autism Spectrum disorder will participate in the Sensory Challenge Protocol which will measure electrodermal activity in response to sensation.
  Interventions: Other: Sensory Challenge Protocol
- Typically Developing Children: typically developing boys between the age of 4 to 11 years will participate in the Sensory Challenge Protocol which will measure electrodermal activity in response to sensation.
  Interventions: Other: Sensory Challenge Protocol

INTERVENTIONS:
Other: Sensory Challenge Protocol — Measurement of electrodermal activity in response to sensation

SUMMARY:
The purpose of this study is tTho establish test-retest reliability of electrodermal markers used to quantify physiologic response to sensation using the Sensory Challenge Protocol in children with and without Autism Spectrum Disorder (ASD).

DETAILED DESCRIPTION:
This methodological research design is a prospective exploratory test-retest design assessing the use of electrodermal activity (EDA) as an index of sensory processing. EDA will be measured using skin conductance response (SCR). The purpose of this study is to investigate if using EDA is a reliable measure over time within the context of response to sensation. Scores from test one and test two of each subject will be correlated to determine reliability of EDA measure. Reliability in this context will establish the utility of EDA as an index of sensory processing. Testing will occur two times within a six week period.

ELIGIBILITY:
Inclusion Criteria: Boys ages 4 - 11 years old.

* Able to sit for 30 minutes and follow simple directions.
* Children with confirmed Autism Spectrum Disorder via school records or parent report.
* Typically developing children free of medical or neurological conditions

Exclusion Criteria:

* Medical or neurological conditions other than Autism.
* Hearing loss or visual impairments.
* Children taking medications known to affect arousal.
* Children who are not able to follow simple commands.

Ages: 4 Years to 11 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A convenience sample of boys between the ages of 4 - 11 years with and without a diagnosis of Autism Spectrum Disorder were recruited from private and public New Jersey Schools, Barpak Occupational Therapy clinic, Bergenfield, New Jersey and Seton Hall University campus.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Electrodermal Activity in response to sensation | within six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barbara M Schupak, PhD, Principal Investigator — Barpak GHS, Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McIntosh DN, Miller LJ, Shyu V, Hagerman RJ. Sensory-modulation disruption, electrodermal responses, and functional behaviors. Dev Med Child Neurol. 1999 Sep;41(9):608-15. doi: 10.1017/s0012162299001267. PMID 10503919
- [Background] Miller LJ, Coll JR, Schoen SA. A randomized controlled pilot study of the effectiveness of occupational therapy for children with sensory modulation disorder. Am J Occup Ther. 2007 Mar-Apr;61(2):228-38. doi: 10.5014/ajot.61.2.228. PMID 17436845
- [Background] Miller LJ, McIntosh DN, McGrath J, Shyu V, Lampe M, Taylor AK, Tassone F, Neitzel K, Stackhouse T, Hagerman RJ. Electrodermal responses to sensory stimuli in individuals with fragile X syndrome: a preliminary report. Am J Med Genet. 1999 Apr 2;83(4):268-79. PMID 10208160
- [Background] Schoen S, Miller LJ, Brett-Green B, Hepburn S. Psychophysiology of children with ASD. Research in Autism Spectrum Disorders 2: 417-429, 2008